CLINICAL TRIAL: NCT04736823
Title: A Phase II Trial of AK112 (PD1/VEGF Bispecific) in Combination With Chemotherapy in Patients With NSCLC
Brief Title: A Trial of AK112 (PD1/VEGF Bispecific) in Combination With Chemotherapy in Patients With NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-201
Record Dates: First submitted 2021-01-30; First posted 2021-02-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed; Paclitaxel; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part1 Cohort1(AK112 + Pemetrexed or Paclitaxel+Carboplatin) (Experimental): non-Squamous NSCLC:Subjects receive AK112 plus Pemetrexed and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK112 plus Pemetrexed until progression.
  Squamous NSCLC:Subjects receive AK112 plus Paclitaxel and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK112 until progression.
  Interventions: Drug: AK112; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin
- Part1 Cohort2(AK112 + Pemetrexed +Carboplatin) (Experimental): Subjects receive AK112 plus Pemetrexed and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK112 plus Pemetrexed until progression.
  Interventions: Drug: AK112; Drug: Pemetrexed; Drug: Carboplatin
- Part1 Cohort3(AK112 + Docetaxel) (Experimental): Subjects receive AK112 plus Docetaxel on Day 1 of every 3-week cycle (Q3W) until progression.
  Interventions: Drug: AK112; Drug: Docetaxel
- Part2 (AK112 + Pemetrexed or Paclitaxel+Carboplatin) (Experimental): non-Squamous NSCLC:Subjects receive AK112 plus Pemetrexed and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK112 plus Pemetrexed until progression.
  Squamous NSCLC:Subjects receive AK112 plus Paclitaxel and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK112 until progression.
  Interventions: Drug: AK112; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin
- Part3 group A(AK112 + Docetaxel) (Experimental): Subjects receive AK112 plus Docetaxel on Day 1 of every 3-week cycle (Q3W) until progression.
  Interventions: Drug: AK112; Drug: Docetaxel
- Part3 group B(AK112) (Experimental): Subjects receive AK112 on Day 1 of every 3-week cycle (Q3W) until progression.
  Interventions: Drug: AK112
- Part3 group C(Docetaxel) (Experimental): Subjects receive Docetaxel on Day 1 of every 3-week cycle (Q3W) until progression.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: AK112 — IV infusion
  Arms: Part1 Cohort1(AK112 + Pemetrexed or Paclitaxel+Carboplatin); Part1 Cohort2(AK112 + Pemetrexed +Carboplatin); Part1 Cohort3(AK112 + Docetaxel); Part2 (AK112 + Pemetrexed or Paclitaxel+Carboplatin); Part3 group A(AK112 + Docetaxel); Part3 group B(AK112)
Drug: Pemetrexed — IV infusion
  Arms: Part1 Cohort1(AK112 + Pemetrexed or Paclitaxel+Carboplatin); Part1 Cohort2(AK112 + Pemetrexed +Carboplatin); Part2 (AK112 + Pemetrexed or Paclitaxel+Carboplatin)
Drug: Paclitaxel — IV infusion
  Arms: Part1 Cohort1(AK112 + Pemetrexed or Paclitaxel+Carboplatin); Part2 (AK112 + Pemetrexed or Paclitaxel+Carboplatin)
Drug: Carboplatin — IV infusion
  Arms: Part1 Cohort1(AK112 + Pemetrexed or Paclitaxel+Carboplatin); Part1 Cohort2(AK112 + Pemetrexed +Carboplatin); Part2 (AK112 + Pemetrexed or Paclitaxel+Carboplatin)
Drug: Docetaxel — IV infusion
  Arms: Part1 Cohort3(AK112 + Docetaxel); Part3 group A(AK112 + Docetaxel); Part3 group C(Docetaxel)

SUMMARY:
This is a phase II study. All patients are stage IIIB/C or IV non-small cell lung cancer(NSCLC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of AK112 in combination with chemotherapy in patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (at the time of inform consent obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Have histologically- or cytologically-confirmed diagnosis of Stage IIIB/C or IV NSCLC.
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy.
* Have a life expectancy of at least 3 months.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator
* Has adequate organ function
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Is currently participating in a study of an investigational agent or using an investigational device;
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment;
* Has undergone major surgery within 30 days prior to the first dose of study treatment;
* Has a known history of prior malignancy except that basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases;
* Has carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study;
* Has an active infection requiring systemic therapy;
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment;
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator;
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Has received a live virus vaccine within 30 days prior to first dose of study treatment
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to approximately 2 years
  ORR is the proportion of subjects with CR or PR , based on RECIST v1.1.

SECONDARY OUTCOMES:
PFS | Up to approximately 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
OS | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.
Disease control rate | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guanzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao Y, Chen G, Chen J, Zhuang L, Du Y, Yu Q, Zhuang W, Zhao Y, Zhou M, Zhang W, Zhang Y, Wan Y, Li W, Song W, Wang ZM, Li B, Xia M, Yang Y, Fang W, Huang Y, Zhang L. AK112, a novel PD-1/VEGF bispecific antibody, in combination with chemotherapy in patients with advanced non-small cell lung cancer (NSCLC): an open-label, multicenter, phase II trial. EClinicalMedicine. 2023 Aug 3;62:102106. doi: 10.1016/j.eclinm.2023.102106. eCollection 2023 Aug. PMID 37593227